CLINICAL TRIAL: NCT04542798
Title: Central Sensitization and Aberrant Nerve Sprouting Possible Explanations for RFA Failure of MBDR in CLBP of FJ Origin: CRF Versus WCRF or PRF-DRG Randomized Clinical Trial
Brief Title: CRF vs WCRF or PRF-DRG in CLBP of FJ Origin and RFA Failure of MBDR: Central Sensitization and Aberrant Nerve Sprouting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital General Universitario de Valencia (Other)
Responsible Party: Principal Investigator, Giuseppe Luca Formicola, Principal Investigator, Hospital General Universitario de Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 34831
Record Dates: First submitted 2020-08-27; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Low Back Pain, Recurrent; Neuropathic Pain; Facet Joint Pain; Central Sensitisation; Aberrant Neuronal Branching; Nociceptive Pain; Mechanical Low Back Pain
Keywords: PULSED RADIOFREQUENCY; WATER-COOLED RADIOFREQUENCY; CONVENTIONAL RADIOFREQUENCY; CHRONIC LOW BACK PAIN; CENTRAL SENSITIZATION; ABERRANT NERVE SPROUTING; FACET JOINT; NEUROPATHIC PAIN; NOCICEPTIVE/MECHANICAL LOW BACK PAIN; RADIOFREQUENCY OF MEDIAL BRANCH OF DORSAL NERVE FAILURE
MeSH Terms: conditions — Low Back Pain; Neuralgia; Nociceptive Pain | interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will not be aware of the technique performed and the data will be collected by a physician unaware of the technique applied. Clinical report form will not contain any identifying data of the patient except for the identification number generated at the time of randomization. The follow up visit will be done identifying the patient by its identification number. After the technique performance, to ensure the blind, the patient will follow the planned out of study postprocedural visit, and a different physician, blind to the technique and to the patient identity, will make the follow up planned at 1, 3 and 6 months. The investigator will open the blind only if it is essential for the patients' management in efficacy and security, and if during the check visit there are clinical reason to do so (mostly severe complications related to the techniques applied and necessity for invasive intervention). The monitor can open the blind for intermediate statistical analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- NPPG (neuropatic pain group) PRF (Experimental): Pulsed radiofrequency neuromodulation of dorsal root ganglia
  Interventions: Device: Radiofrequency COSMAN
- NPPG (neuropatic pain group) CRF (Active Comparator): Conventional radiofrequency ablation of the medial branch of the dorsal nerve
  Interventions: Device: Radiofrequency COSMAN
- NMPG (nociceptive/mechanic pain group) WCRF (Experimental): Water cooled radiofrequency of the medial branch of the dorsal nerve
  Interventions: Device: Radiofrequency COSMAN
- NMPG (nociceptive/mechanic pain group) CRF (Active Comparator): Conventional radiofrequency ablation of the medial branch of the dorsal nerve
  Interventions: Device: Radiofrequency COSMAN

INTERVENTIONS:
Device: Radiofrequency COSMAN — Radiofrequency ablation and neuromodulation
  Other Names: Pulsed Radiofrequency; Water Cooled Radiofrequency; Conventional Radiofrequency

SUMMARY:
The investigators will select two study groups from a population of patients with severe chronic low back pain (CLBP) of facet joint (FJ) origin already treated with conventional radiofrequency ablation (CRFA) of the medial branch of the dorsal ramus (MBDR) and that failed to obtain a 50% pain reduction measured through the numerical rate scale (NRS) for at least 3 months. Severe CLBP is considered a value of at least 7 by NRS pain assessment.

The first group will be characterized by a nociceptive/mechanic type of back pain. The second group of study will be characterized by a neuropathic type of back pain. This difference will be established by a DN4 score of at least 4 points (Doleur Neurophatique 4).

The patients in the group with nociceptive/mechanic back pain will be randomly assigned to conventional radiofrequency ablation or to water cooled radiofrequency (WCRF) of the MBDR. The patients in the group with neuropathic back pain will be randomly assigned CRFA of MBDR or to pulsed radiofrequency (PRF) of the dorsal root ganglia (DRG).

The study will be carried on for an estimated time of 3 years.

Primary outcomes will be:

* at least 50% back pain reduction for at least 3 months evaluated through NRS, with a subcategorization of results that will consider a mean difference in effect (respect to the initial evaluation, with an initial NRS score of at least 7) of 1 point on NRS pain scale as small/modest, 2 points as moderate, more than 2 as large/substantial between the case/control study groups.
* improvement of low back pain disability: 10 points increase on the Oswestry Low Back Pain Disability Questionnaire (ODI) have been proposed as minimal clinically important differences, between 10 and 20 as moderate, more than 20 as large/substantial clinical improvement at month 3 and 6.

Secondary outcome will be evaluated by the 12-item short form survey SF12, accordingly with the clinical pre-interventional findings, analgesic intake at month 1-3-6 (if increased, unchanged, decreased, in dosages or number of pain killers' assumption). Groups sizes: will be calculated based on the disease's incidence and the outcome targets.

DETAILED DESCRIPTION:
The efficacy of radiofrequency to treat LBP of FJ origin decreases with time, and the pathophysiological mechanisms behind this failure is a matter of debate; the phenomenon of central sensitization and ectopic nerve regeneration could be possible explanations.

Central sensitization represents an enhancement in the function of neurons and circuits in nociceptive pathways caused by increases in membrane excitability and synaptic efficacy as well as to reduced inhibition and is a manifestation of the remarkable plasticity of the somatosensory nervous system in response to activity, inflammation, and neural injury. The net effect of central sensitization is to recruit previously subthreshold synaptic inputs to nociceptive neurons, generating an increased or augmented action potential output: a state of facilitation, potentiation, augmentation, or amplification. Central sensitization is responsible for many of the temporal, spatial, and threshold changes in pain sensibility in acute and chronic clinical pain settings and exemplifies the fundamental contribution of the central nervous system to the generation of pain hypersensitivity. Because central sensitization results from changes in the properties of neurons in the central nervous system, the pain is no longer coupled, as acute nociceptive pain is, to the presence, intensity, or duration of noxious peripheral stimuli. Instead, central sensitization produces pain hypersensitivity by changing the sensory response elicited by normal inputs, including those that usually evoke innocuous sensations.

In previous studies using animal models of low back pain, mechanical allodynia has been correlated with and is hypothesized to be due to a host of physiologic changes in the central nervous system. Among these nociceptive responses are neuronal plasticity, glial cell activation and cytokine upregulation. In addition, animal models specifically investigating changes in neural electrical activity following lumbar facet capsule stretching have demonstrated alterations in neurophysiology for applied loading. Together, these molecular and cellular changes contribute to central sensitization and persistent pain. Indeed, in clinical research, central sensitization has been hypothesized as a mechanism of chronic pain after whiplash injury.

Injury to the cervical facet joint and its capsule is primarily a ligamentous injury but because the facet capsule is innervated there may also be neuropathic injury. In fact, capsule stretch in several animal models induces both transient increases in firing of joint-innervating afferents similar to the injury discharge that accompanies nerve injury and also the later development of ectopic firing and hyperexcitability in dorsal horn neurons. The onset of spontaneous firing likely represents a temporal threshold after which sensitization persists despite blockade of joint afferent activity with nerve blocks or neurotomy.

Patients with chronic pain exhibit primary mechanical hyperalgesia over the back of the cervical spine, in a "coat hanger" distribution indicative of peripheral nociceptor sensitization. These patients are also hypersensitive to pressure, heat, and cold stimuli at sites distant from the cervical spine, including over the median, radial, and ulnar nerve trunks in the arm and over the tibialis anterior muscle. Together, these studies demonstrate that generalized and widespread secondary hypersensitivity is robust in individuals who sustain a whiplash-like exposure and indicative of central sensitization. Patient-reported sensory disturbances include spontaneous pain that is disproportionate to and/or occurs in the absence of any inciting event.

There are more than two dozen reported cases of lumbar facet dislocation after rapid deceleration injuries (e.g., traffic accidents), most involving L5-S1. The mechanism of injury in these cases is purported to be a combination of hyperflexion, distraction, and rotation. In a posthumous study conducted in 31 lumbar spines of subjects who died of traumatic injuries (mostly motor vehicle accidents), Twomey et al. found occult bony fractures in the superior articular process or subchondral bone plate in 35% of victims, and z-joint capsular and/or articular cartilage damage in 77% of cases. In this study the authors concluded that occult bony and soft tissue injuries to the l-z joints may be a common cause of LBP after trauma.

In addition to immediate neuronal responses, facet capsular loading that induces behavioural hypersensitivity in the rat is also associated with many sustained modifications in the nociceptive signalling from the primary afferents that are evident in the DRG.

Protein expression of the nociceptive neurotransmitter, substance P, is increased in the DRG after painful facet joint stretch by day 7, and that change is absent in non-painful stretch. Capsular stretch-induced increases in DRG expression of the metabotropic glutamate receptor 5 (mGluR5) and its second messenger, protein kinase C-epsilon (PKCε), are strain dependent and are not evident until 7 days after the initial injury. The late upregulation of these molecules suggests that they may play a role in the later nociceptive pathways involved in injury-induced pain. Because these neuromodulators are involved in neuroplasticity and pain, their delayed elevation implies that the afferents undergo persistent activation and/or dysfunction after painful loading has occurred. Because axonal degeneration is known to take 7 days to develop, it may contribute to the late onset of modified nociceptive signalling.

In addition to increases in expression of glutamate receptors, expression of glutamate transporters on astrocytes and neurons, which regulate the clearance of glutamate away from synapses, like glutamate aspartate transporter, glutamate transporter 1, and excitatory amino-acid carrier 1, is also altered in the spinal cord 1 week after painful facet stretch. While the astrocyte glutamate transporter (glutamate aspartate transporter) is upregulated 1 week after painful injury, both glutamate transporter 1 and excitatory amino-acid carrier 1, which are expressed on other cells, are downregulated, pointing to the widespread and complicated dysregulation of glutamate in pain from facet joint injury.

Like other chronic pain conditions, spinal astrocytes are activated for at least 14 days after painful facet stretch. Mechanical injury to the facet capsule also regulates the production of inflammatory mediators, including proinflammatory cytokines and neurotrophins, in the facet joint itself, as well as in the DRG. Because peripheral inflammation increases hyperexcitability and substance P in DRG neurons, along with pain production, recent studies have begun to elucidate the molecular mechanisms by which peripheral inflammation contributes to central sensitization in the context of facet-mediated pain. Recently, neurotrophins have been implicated both locally in the facet and to be more widespread in the CNS. Nerve growth factor (NGF) increases in the facet joint tissues as early as 1 day after a facet joint distraction that produces pain at that same time. Further, inhibiting NGF signalling also prevents the onset of pain and associated spinal neuron hyperexcitability when anti-NGF is given intra-articularly immediately after capsule stretch and before pain develops, suggesting a critical role of local NGF in initiating pain. Unlike NGF, expression of the neurotrophin brain-derived neurotrophic factor (BDNF) increases in both the DRG and spinal cord at a later time (day 7), with intrathecal administration of the BDNF-sequestering molecule trkB-Fc after facet injury partially reducing pain. Collectively, these NGF and BDNF studies not only reveal important novel pathways emerging as having critical roles in pain from whiplash injury, but also provide potential therapeutic targets for treating joint pain.

Histologic studies have demonstrated that the lumbar facet joints are richly innervated with encapsulated (Ruffini-type endings, Pacinian corpuscles), un-encapsulated, and free nerve endings. The presence of low-threshold, rapidly adapting mechanosensitive neurons suggests that in addition to transmitting nociceptive information, the l-z facet capsule also serves a proprioceptive function. Besides substance P and calcitonin gene-related peptide, a substantial percentage of nerve endings in facet capsules have also been found containing neuropeptide Y, indicating the presence of sympathetic efferent fibers. Nerve fibers have also been found in subchondral bone and intra-articular inclusions of l-z joints, signifying that facet-mediated pain may originate in structures besides the joint capsule. In degenerative lumbar spinal disorders, inflammatory mediators such as prostaglandins and the inflammatory cytokines interleukin 1, interleukin 6, and tumor necrosis factor alpha have been found in facet joint cartilage and synovial tissue.

Wide dynamic range neurons in the dorsal horn may be capable of modulating central sensitization in many chronic pain states. In their study K.P.Quinn et al. comparing painful to non-painful and sham C6/C7 cervical facet joint capsule stretch stimuli in a rat model find out that the proportion of cells in the deep laminae that responded as wide dynamic range neurons was increased in the painful group relative to non-painful or sham groups (p<0.0348).

The significant increase in the number of wide dynamic range neurons classified in the painful group (69% of neurons; p>0.0348) in this study suggests that a phenotypic shift in the response of the neuronal population in the deep laminae of the dorsal horn may play a key role in modulating chronic pain after facet joint injury.

These findings suggest that excessive facet capsule stretch, while not producing visible tearing, can produce functional plasticity of dorsal horn neuronal activity. The increase in neuronal firing across a range of stimulus magnitudes observed at day 7 post-injury that facet-mediated chronic pain following whiplash injury is driven, at least in part, by central sensitization.

Despite the fact that most of the neurophysiological and molecular central and peripheral changes in the low back pain syndrome are related to rat experimental whiplash-like exposure, the investigators consider that the mechanisms of central sensitization related to chronic low back pain of FJ origin can be hypothesised to be the same.

On the other side, the mechanism of aberrant nerve sprouting after previous RFA could explain the necessity to increase the size of the lesion, especially in patients that underwent to multiple treatment with such technique.

Pain recurrence after denervation in medical practice, and nerve regeneration from a third degree nerve injury from different ablation techniques, have a common pathway. This pathway includes macrophage migration, Schwann cell proliferation, CAMs for preparing the basement membrane, NGF on the Schwann cell for axonal sprouting, and increased trophic factors.

Injured axons regenerate at a rate of 1-2 mm/day, although the rate depends on many factors and can vary significantly from individual to individual. Since the length of nerve from the axonal lesion to the lumbar facet joint is approximately 30-40 mm, reinnervation could occur within 3-6 weeks. Regeneration is the primary form of nerve repair when >90% of the axons are injured. In partial nerve injuries when only 20%-30% of the axons are affected, collateral sprouting from preserved axons can contribute to reinnervation. Okuyama et al. showed that radiofrequency ablation in cardiac tissue results in aberrant nerve sprouting within 2 hours after ablation. Therefore, ablation of nerves within the back could have a high likelihood for a similar development, which could cause faster failure rates.

In conclusion this study will select two groups of patients from a population with severe chronic low back pain (CLBP) of facet joint (FJ) origin already treated with conventional radiofrequency ablation (CRFA) of the medial branch of the dorsal rama (MBDR) and that failed to obtain at least a 50% pain reduction measured through the numerical rate scale (NRS). Severe CLBP is considered a patient subjective pain judgement superior to 7 by NRS evaluation.

The first group will be characterized by a nociceptive/mechanic type of back pain. The second group of study will be characterized by a neuropathic type of back pain. This difference will be established by a DN4 score superior to 4 points (Doleur Neurophatique 4) and a negative pre-interventional eco-guided medial branch block (MBB). A negative MBB will be characterized by a reduction of NRS inferior to 50%.

The aim of this study is to try to clarify if a larger lesion created by the water cooled radiofrequency (WCRF) in the nociceptive/mecchanic pain groups (NMPG) and the pulsed radiofrequency (PRF) of dorsal root ganglia (DRG) in the neuropatic pain groups (NPPG) could improve patients' functional status and reduce the burden of their low back pain compared to conventional radiofrequency (CRF) of the medial brach of the dorsal rama (MBDR).

If the hypothesis in study are confirmed there is to be expected a statistically significant reduction in the NRS and an improvement in the ODI score in the DRG-PRF and WCRF groups, compared to the patients in the CRF groups. The aim is to allow the patients to start a program of rehabilitation/physiotherapy, that is by far the standard of clinical care for LBP syndrome.

In this case the results could support our hypothesis in both group of investigations.

Like already underlined in the physiopathological explanation representing the base of this study, increasing the area of lesion with the WCRF technique should increase the chances to target the arborized neural regenerate terminals to the zygapophyseal joint, leading to a better result and possibly longer efficacy of the procedure in the NMPG respect to the group treated with CRF. Today, different doctors use both techniques based on their personal preference and logistic possibility as there are no conclusive data about superiority; even the last consensus practice guidelines for lumbar facet joint pain proposed by the American Society of Regional Anesthesia and Pain Medicine 2020 (CPG-ASRAPM) assess that "there is indirect evidence, and limited direct evidence, that techniques that result in larger lesions (eg, larger electrodes, higher temperatures, longer heating times, proper electrode orientation, fluid modulation) improve outcomes" (Grade C, low level of certainty that larger lesions increase the chance of capturing nerves. Grade I, low level of certainty that larger lesions increase duration of pain relief).

On the other hand, in the NPPG the treatment of the DRG with PRF should interrupts and possibly treat the intercellular and molecular circuits at the base of the central pain sensitization, improving the outcomes considered in this study.

The biggest effort of this study will be the standardization of all the procedures, to allow the maximal reproducibility, in line with the latest recommendation in diagnosis and treatment of low back pain of facet joint origin stated by the CPG-ASRAPM and current best practice in radiofrequency denervation of the lumbar facet joints published by the British Pain Society (CBP-BPS).

The theory that chronic LBP of FJ origin can be related to a central sensitization mechanism is a new investigation field, with no other studies yet exploring our treatment hypothesis.

Therefore, it is important to carry out research projects that clarify which technical variables are those that provide an improvement in pain control and, above all, an improvement in the quality of life in these patients.

Some of the conclusions of this project could be possible applied by professionals of the Pain Units worldwide in their daily activity, in order to provide our patients with the best care and the best possible results. It is a clinical study and therefore its translation to the clinical practice can be direct.

TREATMENTS The application of radiofrequency (RF) signals to neural tissue is well established in the treatment of movement, mood, and chronic pain disorders. Undesired neural signals, such as those transmitting nociceptive pain, are interrupted when high-frequency current (100-1,000 kHz) flowing through an RF probe's active tip raises the temperature at a soma/ganglion or axon/nerve to destructive levels (45-50°C) by means of frictional heating. The process is known as RF heat lesioning, RF thermocoagulation, RF ablation, or thermal RF. The volume of tissue damaged by RF heating is called a heat lesion. Monopolar RF (the technique used in this hospital) refers to current flow between a probe electrode and a large area ground pad placed on the skin's surface. Bipolar RF refers to current flow between two probe electrodes without a ground pad.

RF heat lesioning includes cooled RF, wherein the electrode is internally cooled by circulating fluid but surrounding tissue is exposed to destructive temperatures. Water-cooled radiofrequency (WCRF) ablation is a minimally invasive neuroablative technique used in the treatment of various pain syndromes. The mechanism of pain relief from WC-RF application is analogous to CRF application: a thermal lesion is created, by applying radiofrequency (RF) energy through an electrode placed in the vicinity of the target neural structure, with the aims of interrupting the afferent nociceptive pathways. The difference already mentioned is that the 'cooled' radiofrequency probes have water running through the probe tip, which keeps the tip cooled and allows a larger lesion to be made. Since the physician can't actually see the nerve he is trying to target, larger lesions should theoretically improve his chances of hitting it. The 'cooling' of the water also allows the temperatures to be lower than what is needed for standard RF (approximately 60°C).It is widely accepted that the PRF action mechanism (involving lower temperatures, below 42-44 °C) is most likely related to the induced electric field, rather than to thermal effects. Different effects of exposure to PRF electrical fields have already been reported. Some studies have revealed evidence of morphological changes in the neuronal cells after PRF treatment that affect the inner structures of axons. These structural changes consist of mitochondria swelling and disruption of the normal organisation of the microtubules and microfilaments that preferentially affect C-fibres and to a lesser extent Aδ fibres. In addition, transient ultrastructural changes such as endoneural oedema and collagen deposition have also been found. Besides structural changes, the effects on cellular activity and gene expression have also been observed as well as an increase in the expression of inflammatory proteins. All these effects could potentially inhibit the transmission of nerve signals through C-fibres, which would lead to pain relief.

Number and laterality of medial branches to be lesioned is to be decided after a clinical examination by the pain physician. When selecting targets for blocks, levels should be determined based on clinical presentation, radiological findings when available, tenderness on palpation performed under fluoroscopy. A maximum of eight medial branches at a maximum of four vertebral levels may be lesioned in a single sitting, subjects with unilateral pain to receive unilateral treatment. A maximum of three DRG for each side will be treated in a single sitting.

For various reasons, medial branch blocks are the only acceptable and validated diagnostic test as an indication for medial branch neurotomy. The paradigm of lumbar medial branch neurotomy is that patient's pain can be relieved by coagulating the nerves that mediate (transmit) their pain. An essential prerequisite, therefore, is that it must be shown that the target nerves are responsible for the patient's pain. This is achieved by controlled diagnostic blocks of the medial branches of the cervical and lumbar dorsal rami that mediate the pain. In order to reduce the likelihood of responses being false positive, controlled blocks are mandatory.

An issue in this sense is represented by the relatively high percentage of false positive MBB for placebo effect (up to 30%) described in the literature (patients that responds positively to the MMB, but that fail or will possibly again fail a sustained benefit after the conventional procedure - control group). On the other side some patients may respond positively to the MBB but presents with a neuropathic back pain, possibly leading to a bias in selection, because in this case the mechanisms involved in the origin of back pain could be both neuropathic and nociceptive/mechanic in nature.

Considering the high percentage of placebo related effect in the false positive group, the only way to exclude this kind of false positive is to perform a placebo-controlled pre-procedural MBB, where the placebo procedures will be difficult to be approved by any ethical committee, due to the relatively safety of this procedures.

For this reasons this investigators decided to exclude patients positive to the MBB but with neuropathic pain and the patients with negative MBB and negative DN4 score.

All the patients recruited in this study have been previously treated in our pain service by experienced interventionists anesthesiologists (this will suppose that the percentage of patients actually positive to the MBB because of previous inefficacy technique should be really low).

Indeed, this study group decided to perform a single MBB with 0.5 mL of levo-bupivacaine 5 mg/mL, that is the consensus preferred solution, under ultrasonographic guidance, in our technical operative room, with needle tip to be positioned on the curvature between the articular process and transverse process.

Three radiofrequency techniques have been in use over the past three decades. The scientific community refers to them by name of continents where each was originally described: European, North American, and Australian.

The technique described by Nath and all. and mentioned like standard of treatment in the last consensus on best practice in RFA of the lumbar facet join by the British Pain Society, similar to the Australian technique, is described as follows: the lumbar spine is visualized and the radiograph beam is adjusted to come from a posterior-lateral aspect to get the best possible view of the curvature of the medial part of the upper border of the transverse process where it ascends to become the ventral-lateral border of the superior articular process. In patients with a hypertrophic superior articular process due to arthritic changes greater lateral rotation can be required. The C-arm is then inclined caudal so that the direction of the radiograph beam is from upwards looking below and somewhat medially along the groove in which the medial branch lies.

A 22 SWG SMK C15 cannula with a 5 mm active tip is introduced along the direction of the radiograph beam, in the so-called "tunnel technique" until bone contact is made with the lower part of the transverse process (L5 and higher). The cannula is then rotated so that the bevel was against the bone allowing the needle to slide up in the groove maintaining contact with the bone surface till the tip was at the upper border and in the centre of the curvature formed by the upper border of the transverse process ascending to form the lateral border of the articular process. The position is then checked in the tunnel view, the postero-lateral view as well as a cephalad view. The lateral view confirms that the cannula is not too far in, encroaching on the foramen.

At the S1 level (L5 dorsal ramus) a similar view is maintained to lay the cannula in the groove between the lower part of the lateral aspect of the superior articular process of S1 and the upper surface of the ala of the sacrum. The tunnel view confirms the position in the groove. The forward advance is checked rotating the C-arm to look from a more lateral aspect to visualize the anterior border of the superior articular process of S1, and then from a more cephalad aspect to visualize the point of the needle in relation to the anterior border of the ala of the sacrum.

About the DRG, the radiological location can be divided into 3 types-the intraspinal, foraminal, and extraforaminal regions; most DRG neurons are of the foraminal type. This position corresponds to the dorsal-cranial quadrant of the intervertebral foramen on the lateral view in fluoroscopy, and the middle of the pedicle column on the anteroposterior (AP) view. However, if the arthritic degenerative changes and foraminal stenosis are severe, positioning the needle to target the DRG on fluoroscopy may be difficult. Accordingly, needle tips can be placed laterally on the side of the corresponding pedicle in the AP view. When the RF needle is close to the target position, the stylet of the RF needle is removed, and the RF probe is inserted. Similar to the Australian technique, the C-arm is placed with a 20-30° lateral tilt on the side to treat, with a slightly caudocephalad tilt, to better visualize the foramen, just under the inferior border of the transvers process, with placement of the needle in tunnel vision. The final position of the RF probe is determined with sensory stimulation (50 Hz), at a voltage below 0.5 V. Proximity of the needle to the DRG is determined by appropriate sensory stimulation with 50 Hz (0.4-0.6 V), when the patient feels a tingling sensation. If the threshold value exceeded 0.5V, the needle is carefully advanced until the patient feels sensory stimulation. Motor stimulation at 2 Hz is used to determine a threshold 1.5-2.0 times greater than the sensory threshold to avoid placement near the anterior nerve root and perform the procedure safely. Contrast injection at the end of the needle tip positioning could represent a further confirmation.

Despite the fact that a curved cannula could increase the size of the lesion, a straight 22-gauge cannula with a 5-mm active tip remains the tool most commonly used for radiofrequency denervation of the facet nerves, and it will be the used cannula in the CRF group and in the DRG-PRF group. A 4-mm active tip 10 cm long 17G cannula will be placed for WCRF.

This group of investigation will adopt a modified Nath technique (using a 5 to 15 degree cephalo-caudal inclination and a needle view similar to that obtained with the advanced Australian technique), for CRF and WCRF ablation of MBDR.

Position of the radiofrequency cannula will be confirmed by fluoroscopy with AP, oblique, and lateral view. Once the cannula(e) position is confirmed, routine motor testing will be carried out with a threshold for lower limb muscle contraction of 2V. Lower limb muscle contractions occurring below the threshold will prompt a repositioning of the RF cannula. Sensory stimulation will be applied when single lesions are anticipated (CRF groups); sensory stimulation of 0,6V mean that the needle is placed at less than 3 mm from the MBDR, that is the ideal distance to realize an adequate lesion. When multiple or large lesions are planned, the evidence for sensory stimulation is inconclusive; despite this fact, it was decided to check for sensory stimulation for all patients involved in this study, knowing that in the WCRF and CRF groups such stimulation could be inconclusive.

Due to the larger expected lesion size in the WCRF, like suggested by the work of Malik et all. the investigators will ensure a "safe distance" from the segmental spinal nerve by adopting the following safety measures: (a) the electrode tip will be placed on the transverse process, about 4 mm lateral to its junction with the superior articular process; (b) the parameters used for sensory testing will be modified and paresthesia will be sought at > 0.6 V, between 0.8 V to 1.0 V.

In the case of CRF and WCRF before starting the treatment, 1 ml of lidocaine 1% will be injected through the cannula.

Each lesion will be carried out at 80° C for 90 seconds in the CRF group. One lesions will be applied for each treated level.

Each lesion in the WCRF group will be carried out at 60° C for 150 seconds. One lesion will be applied for each treated level.

At the end of the procedure 1 to 1.5 ml of a mixture of ropivacaine 0,2% 8ml + betamethasone 11.8 mg 2ml will be injected before the extraction of the needle, in both this groups.

In the case of DRG-PRF, a pulsed current (20ms, 2 Hz) is applied (1 time for 120 seconds), with a 45V output, 20ms lasting impulse (480ms pause). During this procedure, the temperature at the tip of the electrode is not supposed to exceed 42℃.

At the end of the procedure, 0,5 to 1 ml of a mixture of ropivacaine 0,1% 8ml and dexamethasone 8mg will be injected before needle extraction.

The CRF treatment and the DRG-PRF will be realized with the Cosman G4 Radiofrequency Generator. For the WCRF a COOLED RF Generator of Halyard will be used. All the procedures can be performed in day hospital, with no need for hospitalization.

Ones the needle is positioned, the wire is retired and the probe is inserted; the measured impedance has to be between 200 and 700Ω to confirm the proximity to the target structure.

All patients will be in a prone position.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic lumbar back pain supposed to be of facet joint origin (low back pain irradiated to buttocks, legs, eventually feet in absence of exclusion criteria);
* positivity to FJ provocative clinical tests, possible muscle spasm over the affected joints;
* positivity to DN4 assessment in the NPPG + negative MBB and negative DN4 assessment + positive MMB in the NMPG;
* efficacy of MBDR-RF treatment for at least one time reported in the personal clinical history, unresponsive to the last CRF or WCRF (only for the NPPG);
* an MRI no more than 2 years;
* basal NRS ≥ 7;
* patients between 18y and 85y;
* ASA (American Society of Anaesthesiologists scale) I-III;
* absence of severe chronic disease associated, full mental capacity to sign the informed consent.

This group is well aware that nowadays literature lack of confirmed clinical diagnostic criteria, like underlined in the last CPG-ASRAPM. Despite this issue, we decided to select our clinical criteria to better identify LBP of FJ origin following some of the indications mentioned in the Delphi survey of an expert panel (Wilde et al., 2007):

* reproduction of similar or even worsening of basal pain during paravertebral finger pressure applied no more than 2-3 cm laterally to the midline (89% expert acceptance);
* improvement of patient's pain during the flexion of the trunk while sitting (78% expert acceptance);
* reduced range of motion or increased stiffness during local lateral passive movements (61% expert acceptance);
* positive balance test with increased pain during extension - stress movements (after the flexion manoeuvre), or during lateral flexion (starting from 20 degree) and rotational axial movements (56% expert acceptance).
* Another manoeuvre, taking into consideration the spinal columns' biomechanics, is realized asking the patients while standing with joined feet, to flex completely the trunk trying to touch with hands the top of his feet; this movement should not provoke patients' usual pain or worsen it; after that is invited to slowly return to a neutral position, stopping for 5 seconds in a 90-degree position between the trunk and the feet; during the extension movement to recover the initial position, the pain could worsen, or mimic the patients' usual pain, but it can't improve.

We decided to include also patient that present with bilateral low back pain, despite this survey describe localized unilateral low back pain like one of possible clinical indicator of lumbar facet joint pain (80% expert agreement); this decision is based on our clinical experience.

Exclusion Criteria:

* positive MBB with positive DN4;
* negative MMB with negative DN4;
* positive EMG for neuropathic pain of radicular origin (89% expert acceptance),
* diagnostic imaging of significant radicular compression (based on the radiologist judgement);
* late diagnosis of other causes of LBP, cancer related pain, neoplastic patients, patients with life expectation inferior to 1 year;
* BMI > 35;
* patients insurance or work absence related interests
* patient refusal
* Back's depression inventory II (BDI-II) > 20,
* previous lumbar spinal, pelvic and knee surgery, or significant stenosis of the spinal canal that can interfere with diagnosis;
* patient with systemic infection, pregnant or breastfeeding woman, untreatable coagulative problems;
* clinical doubt by the enrolling physician that can interfere with the evaluation's efficacy of the procedures under investigation (like hip pain, cluneal nerve's entrapment pain, trochanteritis, myofascial pain, etc.);
* any contraindication to neuraxial injection.
* Social risk factors that could influence the adherence to the study protocol will be taken into consideration and valuated accordingly.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
PNRS change >= 50% | 3 and 6 months
  At least 50% back pain reduction for at least 3 months valuated through NRS, with a subcategorization of results that will consider a mean difference in effect (respect to the initial evaluation, with a NRS score of at least 7) of 1 point on NRS pain scale as small/modest, 2 points as moderate, more than 2 as large/substantial between the case/control study groups.
ODI change > 10 points | 3 and 6 months
  Improvement of low back pain disability: 10 points reduction on the Oswestry Low Back Pain Disability Questionnaire (ODI) have been proposed as minimal clinically important differences, between 10 and 20 as moderate, more than 20 as large/substantial clinical improvement at month 3 and 6.

SECONDARY OUTCOMES:
SF12 change >= 20 points | 3 and 6 months
  Quality of life improvement valuated through a SF12 questionnaire, with an increase of post-procedural score of at least 20 points.
Pain killer drugs intake | 6 mounths
  Reduced pain drugs intake at month 6 post-procedural. A reduced intake will be considered a reduction of at least 30% of occasional pain killers and a reduction of 30% of opioids dosage intake (if regularly assumed).

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Luca Formicola, MD, Principal Investigator — Fellow at the General Universitary Hospital of Valencia, Department of Pain Medicine, Resident in Anesthesia and Intensive Care of San Raffaele Hospital, Milan, Italy; Gustavo Fabregat Cid, MD, PhD, Principal Investigator — MD, PhD at Multidisciplinary Pain Management Unit, Anesthesia, Critical Care, and Pain Management Department, General University Hospital, Valencia, Spain
Locations (1):
- General Universitary Hospital of Valencia, Valencia, Spain

REFERENCES:
- [Background] Ashton IK, Ashton BA, Gibson SJ, Polak JM, Jaffray DC, Eisenstein SM. Morphological basis for back pain: the demonstration of nerve fibers and neuropeptides in the lumbar facet joint capsule but not in ligamentum flavum. J Orthop Res. 1992 Jan;10(1):72-8. doi: 10.1002/jor.1100100109. PMID 1530799
- [Background] Avramov AI, Cavanaugh JM, Ozaktay CA, Getchell TV, King AI. The effects of controlled mechanical loading on group-II, III, and IV afferent units from the lumbar facet joint and surrounding tissue. An in vitro study. J Bone Joint Surg Am. 1992 Dec;74(10):1464-71. PMID 1469006
- [Background] Back SH, Kowey PR. Strategies to Reduce Recurrent Shocks Due to Ventricular Arrhythmias in Patients with an Implanted Cardioverter-Defibrillator. Arrhythm Electrophysiol Rev. 2019 May;8(2):99-104. doi: 10.15420/aer.2018.55.5. PMID 31114683
- [Background] Barlas P, Walsh DM, Baxter GD, Allen JM. Delayed onset muscle soreness: effect of an ischaemic block upon mechanical allodynia in humans. Pain. 2000 Aug;87(2):221-225. doi: 10.1016/S0304-3959(00)00287-6. PMID 10924815
- [Background] Beaman DN, Graziano GP, Glover RA, Wojtys EM, Chang V. Substance P innervation of lumbar spine facet joints. Spine (Phila Pa 1976). 1993 Jun 15;18(8):1044-9. doi: 10.1097/00007632-199306150-00014. PMID 7690159
- [Background] Bombardier C, Hayden J, Beaton DE. Minimal clinically important difference. Low back pain: outcome measures. J Rheumatol. 2001 Feb;28(2):431-8. PMID 11246692
- [Background] Borchers AT, Gershwin ME. Complex regional pain syndrome: a comprehensive and critical review. Autoimmun Rev. 2014 Mar;13(3):242-65. doi: 10.1016/j.autrev.2013.10.006. Epub 2013 Oct 23. PMID 24161450
- [Background] BRODKEY JS, MIYAZAKI Y, ERVIN FR, MARK VH. REVERSIBLE HEAT LESIONS WITH RADIOFREQUENCY CURRENT. A METHOD OF STEREOTACTIC LOCALIZATION. J Neurosurg. 1964 Jan;21:49-53. doi: 10.3171/jns.1964.21.1.0049. No abstract available. PMID 14110358
- [Background] Cavanaugh JM, Ozaktay AC, Yamashita HT, King AI. Lumbar facet pain: biomechanics, neuroanatomy and neurophysiology. J Biomech. 1996 Sep;29(9):1117-29. doi: 10.1016/0021-9290(96)00023-1. PMID 8872268
- [Background] Chang YW, Winkelstein BA. Schwann cell proliferation and macrophage infiltration are evident at day 14 after painful cervical nerve root compression in the rat. J Neurotrauma. 2011 Dec;28(12):2429-38. doi: 10.1089/neu.2011.1918. Epub 2011 Sep 21. PMID 21787151
- [Background] Chapman JR, Norvell DC, Hermsmeyer JT, Bransford RJ, DeVine J, McGirt MJ, Lee MJ. Evaluating common outcomes for measuring treatment success for chronic low back pain. Spine (Phila Pa 1976). 2011 Oct 1;36(21 Suppl):S54-68. doi: 10.1097/BRS.0b013e31822ef74d. PMID 21952190
- [Background] Chen C, Lu Y, Kallakuri S, Patwardhan A, Cavanaugh JM. Distribution of A-delta and C-fiber receptors in the cervical facet joint capsule and their response to stretch. J Bone Joint Surg Am. 2006 Aug;88(8):1807-16. doi: 10.2106/JBJS.E.00880. PMID 16882906
- [Background] Cheng J, Pope JE, Dalton JE, Cheng O, Bensitel A. Comparative outcomes of cooled versus traditional radiofrequency ablation of the lateral branches for sacroiliac joint pain. Clin J Pain. 2013 Feb;29(2):132-7. doi: 10.1097/AJP.0b013e3182490a17. PMID 22688606
- [Background] Choi EJ, Choi YM, Jang EJ, Kim JY, Kim TK, Kim KH. Neural Ablation and Regeneration in Pain Practice. Korean J Pain. 2016 Jan;29(1):3-11. doi: 10.3344/kjp.2016.29.1.3. Epub 2016 Jan 4. PMID 26839664
- [Background] Choi S, Choi HJ, Cheong Y, Chung SH, Park HK, Lim YJ. Inflammatory responses and morphological changes of radiofrequency-induced rat sciatic nerve fibres. Eur J Pain. 2014 Feb;18(2):192-203. doi: 10.1002/j.1532-2149.2013.00391.x. Epub 2013 Aug 23. PMID 24038618
- [Background] Chou R, Qaseem A, Owens DK, Shekelle P; Clinical Guidelines Committee of the American College of Physicians. Diagnostic imaging for low back pain: advice for high-value health care from the American College of Physicians. Ann Intern Med. 2011 Feb 1;154(3):181-9. doi: 10.7326/0003-4819-154-3-201102010-00008. PMID 21282698
- [Background] Christensen MD, Hulsebosch CE. Chronic central pain after spinal cord injury. J Neurotrauma. 1997 Aug;14(8):517-37. doi: 10.1089/neu.1997.14.517. PMID 9300563
- [Background] Claycomb KI, Johnson KM, Winokur PN, Sacino AV, Crocker SJ. Astrocyte regulation of CNS inflammation and remyelination. Brain Sci. 2013 Jul 22;3(3):1109-27. doi: 10.3390/brainsci3031109. PMID 24961523
- [Background] Coghill RC, Mayer DJ, Price DD. The roles of spatial recruitment and discharge frequency in spinal cord coding of pain: a combined electrophysiological and imaging investigation. Pain. 1993 Jun;53(3):295-309. doi: 10.1016/0304-3959(93)90226-F. PMID 8351159
- [Background] Cohen SP, Bhaskar A, Bhatia A, Buvanendran A, Deer T, Garg S, Hooten WM, Hurley RW, Kennedy DJ, McLean BC, Moon JY, Narouze S, Pangarkar S, Provenzano DA, Rauck R, Sitzman BT, Smuck M, van Zundert J, Vorenkamp K, Wallace MS, Zhao Z. Consensus practice guidelines on interventions for lumbar facet joint pain from a multispecialty, international working group. Reg Anesth Pain Med. 2020 Jun;45(6):424-467. doi: 10.1136/rapm-2019-101243. Epub 2020 Apr 3. PMID 32245841
- [Background] Cohen SP, Hurley RW, Buckenmaier CC 3rd, Kurihara C, Morlando B, Dragovich A. Randomized placebo-controlled study evaluating lateral branch radiofrequency denervation for sacroiliac joint pain. Anesthesiology. 2008 Aug;109(2):279-88. doi: 10.1097/ALN.0b013e31817f4c7c. PMID 18648237
- [Background] Cosman ER Jr, Dolensky JR, Hoffman RA. Factors that affect radiofrequency heat lesion size. Pain Med. 2014 Dec;15(12):2020-36. doi: 10.1111/pme.12566. Epub 2014 Oct 14. PMID 25312825
- [Background] Crosby ND, Gilliland TM, Winkelstein BA. Early afferent activity from the facet joint after painful trauma to its capsule potentiates neuronal excitability and glutamate signaling in the spinal cord. Pain. 2014 Sep;155(9):1878-1887. doi: 10.1016/j.pain.2014.06.019. Epub 2014 Jun 28. PMID 24978827
- [Background] Crosby ND, Weisshaar CL, Winkelstein BA. Spinal neuronal plasticity is evident within 1 day after a painful cervical facet joint injury. Neurosci Lett. 2013 May 10;542:102-6. doi: 10.1016/j.neulet.2013.03.019. Epub 2013 Mar 21. PMID 23523644
- [Background] Curatolo M, Petersen-Felix S, Arendt-Nielsen L, Giani C, Zbinden AM, Radanov BP. Central hypersensitivity in chronic pain after whiplash injury. Clin J Pain. 2001 Dec;17(4):306-15. doi: 10.1097/00002508-200112000-00004. PMID 11783810
- [Background] Das De S, McCreath SW. Lumbosacral fracture-dislocations. A report of four cases. J Bone Joint Surg Br. 1981 Feb;63-B(1):58-60. doi: 10.1302/0301-620X.63B1.7225186.
- [Background] Datta S, Lee M, Falco FJ, Bryce DA, Hayek SM. Systematic assessment of diagnostic accuracy and therapeutic utility of lumbar facet joint interventions. Pain Physician. 2009 Mar-Apr;12(2):437-60. PMID 19305489
- [Background] DeLeo JA, Yezierski RP. The role of neuroinflammation and neuroimmune activation in persistent pain. Pain. 2001 Feb 1;90(1-2):1-6. doi: 10.1016/s0304-3959(00)00490-5. No abstract available. PMID 11166964
- [Background] Deyo RA, Weinstein JN. Low back pain. N Engl J Med. 2001 Feb 1;344(5):363-70. doi: 10.1056/NEJM200102013440508. No abstract available. PMID 11172169
- [Background] Dieckmann G, Gabriel E, Hassler R. Size, form and structural peculiarities of experimental brailesions obtained by thermocontrolled radiofrequency. Confin Neurol. 1965;26(3):134-42. doi: 10.1159/000104015. No abstract available. PMID 4957778
- [Background] Dong L, Quindlen JC, Lipschutz DE, Winkelstein BA. Whiplash-like facet joint loading initiates glutamatergic responses in the DRG and spinal cord associated with behavioral hypersensitivity. Brain Res. 2012 Jun 21;1461:51-63. doi: 10.1016/j.brainres.2012.04.026. Epub 2012 Apr 21. PMID 22578356
- [Background] Dong L, Winkelstein BA. Simulated whiplash modulates expression of the glutamatergic system in the spinal cord suggesting spinal plasticity is associated with painful dynamic cervical facet loading. J Neurotrauma. 2010 Jan;27(1):163-74. doi: 10.1089/neu.2009.0999. PMID 19772459
- [Background] Dreyfuss P, Halbrook B, Pauza K, Joshi A, McLarty J, Bogduk N. Efficacy and validity of radiofrequency neurotomy for chronic lumbar zygapophysial joint pain. Spine (Phila Pa 1976). 2000 May 15;25(10):1270-7. doi: 10.1097/00007632-200005150-00012. PMID 10806505
- [Background] el-Bohy A, Cavanaugh JM, Getchell ML, Bulas T, Getchell TV, King AI. Localization of substance P and neurofilament immunoreactive fibers in the lumbar facet joint capsule and supraspinous ligament of the rabbit. Brain Res. 1988 Sep 20;460(2):379-82. doi: 10.1016/0006-8993(88)90386-1. PMID 2465064
- [Background] Eldabe S, Tariq A, Nath S, Gulve A, Antrobus H, Baloch M, Buczkowski P, Collighan N, Fernandez T, Fritz AK, Humble S, Huygen F, Krishnan M, Mehta V, Mishra S, Muthukrishnan S, Snidvongs S, Tamosauskas R, Underwood M. Best practice in radiofrequency denervation of the lumbar facet joints: a consensus technique. Br J Pain. 2020 Feb;14(1):47-56. doi: 10.1177/2049463719840053. Epub 2019 Apr 3. PMID 32110398
- [Background] Erdine S, Bilir A, Cosman ER, Cosman ER Jr. Ultrastructural changes in axons following exposure to pulsed radiofrequency fields. Pain Pract. 2009 Nov-Dec;9(6):407-17. doi: 10.1111/j.1533-2500.2009.00317.x. Epub 2009 Sep 15. PMID 19761513
- [Background] Frohling MA, Schlote W, Wolburg-Buchholz K. Nonselective nerve fibre damage in peripheral nerves after experimental thermocoagulation. Acta Neurochir (Wien). 1998;140(12):1297-302. doi: 10.1007/s007010050253. PMID 9932132
- [Background] Giles LG. Human lumbar zygapophyseal joint inferior recess synovial folds: a light microscope examination. Anat Rec. 1988 Feb;220(2):117-24. doi: 10.1002/ar.1092200202. PMID 2451453
- [Background] Giles LG, Taylor JR. Innervation of lumbar zygapophyseal joint synovial folds. Acta Orthop Scand. 1987 Feb;58(1):43-6. doi: 10.3109/17453678709146341. PMID 2437759
- [Background] Goldberg SN, Gazelle GS, Solbiati L, Rittman WJ, Mueller PR. Radiofrequency tissue ablation: increased lesion diameter with a perfusion electrode. Acad Radiol. 1996 Aug;3(8):636-44. doi: 10.1016/s1076-6332(96)80188-7. PMID 8796727
- [Background] Goldberg SN, Solbiati L, Hahn PF, Cosman E, Conrad JE, Fogle R, Gazelle GS. Large-volume tissue ablation with radio frequency by using a clustered, internally cooled electrode technique: laboratory and clinical experience in liver metastases. Radiology. 1998 Nov;209(2):371-9. doi: 10.1148/radiology.209.2.9807561.
- [Background] Hains BC, Johnson KM, Eaton MJ, Willis WD, Hulsebosch CE. Serotonergic neural precursor cell grafts attenuate bilateral hyperexcitability of dorsal horn neurons after spinal hemisection in rat. Neuroscience. 2003;116(4):1097-110. doi: 10.1016/s0306-4522(02)00729-7. PMID 12617951
- [Background] Hao JX, Xu XJ, Yu YX, Seiger A, Wiesenfeld-Hallin Z. Transient spinal cord ischemia induces temporary hypersensitivity of dorsal horn wide dynamic range neurons to myelinated, but not unmyelinated, fiber input. J Neurophysiol. 1992 Aug;68(2):384-91. doi: 10.1152/jn.1992.68.2.384. PMID 1527565
- [Background] Hartvigsen J, Hancock MJ, Kongsted A, Louw Q, Ferreira ML, Genevay S, Hoy D, Karppinen J, Pransky G, Sieper J, Smeets RJ, Underwood M; Lancet Low Back Pain Series Working Group. What low back pain is and why we need to pay attention. Lancet. 2018 Jun 9;391(10137):2356-2367. doi: 10.1016/S0140-6736(18)30480-X. Epub 2018 Mar 21. PMID 29573870
- [Background] Heavner JE, Boswell MV, Racz GB. A comparison of pulsed radiofrequency and continuous radiofrequency on thermocoagulation of egg white in vitro. Pain Physician. 2006 Apr;9(2):135-7. PMID 16703974
- [Background] Herrero JF, Headley MP. The dominant class of somatosensory neurone recorded in the spinal dorsal horn of awake sheep has wide dynamic range properties. Pain. 1995 Apr;61(1):133-138. doi: 10.1016/0304-3959(94)00152-5. PMID 7644236
- [Background] Hubbard RD, Quinn KP, Martinez JJ, Winkelstein BA. The role of graded nerve root compression on axonal damage, neuropeptide changes, and pain-related behaviors. Stapp Car Crash J. 2008 Nov;52:33-58. doi: 10.4271/2008-22-0002. PMID 19085157
- [Background] Igarashi A, Kikuchi S, Konno S, Olmarker K. Inflammatory cytokines released from the facet joint tissue in degenerative lumbar spinal disorders. Spine (Phila Pa 1976). 2004 Oct 1;29(19):2091-5. doi: 10.1097/01.brs.0000141265.55411.30. PMID 15454697
- [Background] Ita ME, Zhang S, Holsgrove TP, Kartha S, Winkelstein BA. The Physiological Basis of Cervical Facet-Mediated Persistent Pain: Basic Science and Clinical Challenges. J Orthop Sports Phys Ther. 2017 Jul;47(7):450-461. doi: 10.2519/jospt.2017.7255. Epub 2017 Jun 16. PMID 28622486
- [Background] Jarvik JG, Deyo RA. Diagnostic evaluation of low back pain with emphasis on imaging. Ann Intern Med. 2002 Oct 1;137(7):586-97. doi: 10.7326/0003-4819-137-7-200210010-00010. PMID 12353946
- [Background] Ji RR, Woolf CJ. Neuronal plasticity and signal transduction in nociceptive neurons: implications for the initiation and maintenance of pathological pain. Neurobiol Dis. 2001 Feb;8(1):1-10. doi: 10.1006/nbdi.2000.0360. PMID 11162235
- [Background] Kallakuri S, Singh A, Lu Y, Chen C, Patwardhan A, Cavanaugh JM. Tensile stretching of cervical facet joint capsule and related axonal changes. Eur Spine J. 2008 Apr;17(4):556-63. doi: 10.1007/s00586-007-0562-0. Epub 2007 Dec 14. PMID 18080147
- [Background] Kim WJ, Park HS, Park MK. The effect of needle tip position on the analgesic efficacy of pulsed radiofrequency treatment in patients with chronic lumbar radicular pain: a retrospective observational study. Korean J Pain. 2019 Oct 1;32(4):280-285. doi: 10.3344/kjp.2019.32.4.280. PMID 31569920
- [Background] Kivioja J, Rinaldi L, Ozenci V, Kouwenhoven M, Kostulas N, Lindgren U, Link H. Chemokines and their receptors in whiplash injury: elevated RANTES and CCR-5. J Clin Immunol. 2001 Jul;21(4):272-7. doi: 10.1023/a:1010931309088. PMID 11506197
- [Background] Kovacs FM, Abraira V, Royuela A, Corcoll J, Alegre L, Cano A, Muriel A, Zamora J, del Real MT, Gestoso M, Mufraggi N. Minimal clinically important change for pain intensity and disability in patients with nonspecific low back pain. Spine (Phila Pa 1976). 2007 Dec 1;32(25):2915-20. doi: 10.1097/BRS.0b013e31815b75ae. PMID 18246018
- [Background] Kras JV, Kartha S, Winkelstein BA. Intra-articular nerve growth factor regulates development, but not maintenance, of injury-induced facet joint pain & spinal neuronal hypersensitivity. Osteoarthritis Cartilage. 2015 Nov;23(11):1999-2008. doi: 10.1016/j.joca.2015.06.012. PMID 26521746
- [Background] Kras JV, Tanaka K, Gilliland TM, Winkelstein BA. An anatomical and immunohistochemical characterization of afferents innervating the C6-C7 facet joint after painful joint loading in the rat. Spine (Phila Pa 1976). 2013 Mar 15;38(6):E325-31. doi: 10.1097/BRS.0b013e318285b5bb. PMID 23324931
- [Background] Kras JV, Weisshaar CL, Quindlen J, Winkelstein BA. Brain-derived neurotrophic factor is upregulated in the cervical dorsal root ganglia and spinal cord and contributes to the maintenance of pain from facet joint injury in the rat. J Neurosci Res. 2013 Oct;91(10):1312-21. doi: 10.1002/jnr.23254. Epub 2013 Aug 6. PMID 23918351
- [Background] Lambeek LC, van Tulder MW, Swinkels IC, Koppes LL, Anema JR, van Mechelen W. The trend in total cost of back pain in The Netherlands in the period 2002 to 2007. Spine (Phila Pa 1976). 2011 Jun;36(13):1050-8. doi: 10.1097/BRS.0b013e3181e70488. PMID 21150697
- [Background] Lee KE, Davis MB, Winkelstein BA. Capsular ligament involvement in the development of mechanical hyperalgesia after facet joint loading: behavioral and inflammatory outcomes in a rodent model of pain. J Neurotrauma. 2008 Nov;25(11):1383-93. doi: 10.1089/neu.2008.0700. PMID 19061382
- [Background] Lee KE, Winkelstein BA. Joint distraction magnitude is associated with different behavioral outcomes and substance P levels for cervical facet joint loading in the rat. J Pain. 2009 Apr;10(4):436-45. doi: 10.1016/j.jpain.2008.11.009. PMID 19327645
- [Background] Lord SM, Barnsley L, Wallis BJ, McDonald GJ, Bogduk N. Percutaneous radio-frequency neurotomy for chronic cervical zygapophyseal-joint pain. N Engl J Med. 1996 Dec 5;335(23):1721-6. doi: 10.1056/NEJM199612053352302. PMID 8929263
- [Background] Robinson LR. Traumatic injury to peripheral nerves. Muscle Nerve. 2000 Jun;23(6):863-73. doi: 10.1002/(sici)1097-4598(200006)23:63.0.co;2-0. PMID 10842261
- [Background] Lu Y, Chen C, Kallakuri S, Patwardhan A, Cavanaugh JM. Neural response of cervical facet joint capsule to stretch: a study of whiplash pain mechanism. Stapp Car Crash J. 2005 Nov;49:49-65. doi: 10.4271/2005-22-0003. PMID 17096268
- [Background] Malik K, Benzon HT, Walega D. Water-cooled radiofrequency: a neuroablative or a neuromodulatory modality with broader applications? Case Rep Anesthesiol. 2011;2011:263101. doi: 10.1155/2011/263101. Epub 2011 Dec 18. PMID 22606384
- [Background] Manchikanti L, Singh V, Falco FJ, Cash KM, Fellows B. Cervical medial branch blocks for chronic cervical facet joint pain: a randomized, double-blind, controlled trial with one-year follow-up. Spine (Phila Pa 1976). 2008 Aug 1;33(17):1813-20. doi: 10.1097/BRS.0b013e31817b8f88. PMID 18670333
- [Background] McCarty TR, Garg R, Rustagi T. Efficacy and safety of radiofrequency ablation for treatment of chronic radiation proctitis: A systematic review and meta-analysis. J Gastroenterol Hepatol. 2019 Sep;34(9):1479-1485. doi: 10.1111/jgh.14729. Epub 2019 Jul 2. PMID 31111527
- [Background] McCormick ZL, Choi H, Reddy R, Syed RH, Bhave M, Kendall MC, Khan D, Nagpal G, Teramoto M, Walega DR. Randomized prospective trial of cooled versus traditional radiofrequency ablation of the medial branch nerves for the treatment of lumbar facet joint pain. Reg Anesth Pain Med. 2019 Mar;44(3):389-397. doi: 10.1136/rapm-2018-000035. PMID 30777903
- [Background] McLain RF. Mechanoreceptor endings in human cervical facet joints. Spine (Phila Pa 1976). 1994 Mar 1;19(5):495-501. doi: 10.1097/00007632-199403000-00001. PMID 8184340
- [Background] Goldberg SN, Gazelle GS, Dawson SL, Rittman WJ, Mueller PR, Rosenthal DI. Tissue ablation with radiofrequency: effect of probe size, gauge, duration, and temperature on lesion volume. Acad Radiol. 1995 May;2(5):399-404. doi: 10.1016/s1076-6332(05)80342-3. PMID 9419582
- [Background] Nath S, Nath CA, Pettersson K. Percutaneous lumbar zygapophysial (Facet) joint neurotomy using radiofrequency current, in the management of chronic low back pain: a randomized double-blind trial. Spine (Phila Pa 1976). 2008 May 20;33(12):1291-7; discussion 1298. doi: 10.1097/BRS.0b013e31817329f0. PMID 18496338
- [Background] Okuyama Y, Pak HN, Miyauchi Y, Liu YB, Chou CC, Hayashi H, Fu KJ, Kerwin WF, Kar S, Hata C, Karagueuzian HS, Fishbein MC, Chen PS, Chen LS. Nerve sprouting induced by radiofrequency catheter ablation in dogs. Heart Rhythm. 2004 Dec;1(6):712-7. doi: 10.1016/j.hrthm.2004.09.012. PMID 15851243
- [Background] Ostelo RW, de Vet HC. Clinically important outcomes in low back pain. Best Pract Res Clin Rheumatol. 2005 Aug;19(4):593-607. doi: 10.1016/j.berh.2005.03.003. PMID 15949778
- [Background] Perolat R, Kastler A, Nicot B, Pellat JM, Tahon F, Attye A, Heck O, Boubagra K, Grand S, Krainik A. Facet joint syndrome: from diagnosis to interventional management. Insights Imaging. 2018 Oct;9(5):773-789. doi: 10.1007/s13244-018-0638-x. Epub 2018 Aug 8. PMID 30090998
- [Background] Picavet HS, Schouten JS. Musculoskeletal pain in the Netherlands: prevalences, consequences and risk groups, the DMC(3)-study. Pain. 2003 Mar;102(1-2):167-78. doi: 10.1016/s0304-3959(02)00372-x. PMID 12620608
- [Background] Pinski SE, King KB, Davidson BS, Zhou BH, Lu Y, Solomonow M. High-frequency loading of lumbar ligaments increases proinflammatory cytokines expression in a feline model of repetitive musculoskeletal disorder. Spine J. 2010 Dec;10(12):1078-85. doi: 10.1016/j.spinee.2010.08.030. Epub 2010 Oct 12. PMID 20933478
- [Background] Podhajsky RJ, Sekiguchi Y, Kikuchi S, Myers RR. The histologic effects of pulsed and continuous radiofrequency lesions at 42 degrees C to rat dorsal root ganglion and sciatic nerve. Spine (Phila Pa 1976). 2005 May 1;30(9):1008-13. doi: 10.1097/01.brs.0000161005.31398.58. PMID 15864151
- [Background] Protasoni M, Reguzzoni M, Sangiorgi S, Reverberi C, Borsani E, Rodella LF, Dario A, Tomei G, Dell'Orbo C. Pulsed radiofrequency effects on the lumbar ganglion of the rat dorsal root: a morphological light and transmission electron microscopy study at acute stage. Eur Spine J. 2009 Apr;18(4):473-8. doi: 10.1007/s00586-008-0870-z. Epub 2009 Jan 27. PMID 19172311
- [Background] Quinn KP, Dong L, Golder FJ, Winkelstein BA. Neuronal hyperexcitability in the dorsal horn after painful facet joint injury. Pain. 2010 Nov;151(2):414-421. doi: 10.1016/j.pain.2010.07.034. Epub 2010 Aug 23. PMID 20739124
- [Background] Chou R, Qaseem A, Snow V, Casey D, Cross JT Jr, Shekelle P, Owens DK; Clinical Efficacy Assessment Subcommittee of the American College of Physicians; American College of Physicians; American Pain Society Low Back Pain Guidelines Panel. Diagnosis and treatment of low back pain: a joint clinical practice guideline from the American College of Physicians and the American Pain Society. Ann Intern Med. 2007 Oct 2;147(7):478-91. doi: 10.7326/0003-4819-147-7-200710020-00006. PMID 17909209
- [Background] Ramer MS, French GD, Bisby MA. Wallerian degeneration is required for both neuropathic pain and sympathetic sprouting into the DRG. Pain. 1997 Aug;72(1-2):71-8. doi: 10.1016/s0304-3959(97)00019-5. PMID 9272789
- [Background] Rutkowski MD, Winkelstein BA, Hickey WF, Pahl JL, DeLeo JA. Lumbar nerve root injury induces central nervous system neuroimmune activation and neuroinflammation in the rat: relationship to painful radiculopathy. Spine (Phila Pa 1976). 2002 Aug 1;27(15):1604-13. doi: 10.1097/00007632-200208010-00003. PMID 12163719
- [Background] Sandkuhler J. Learning and memory in pain pathways. Pain. 2000 Nov;88(2):113-118. doi: 10.1016/S0304-3959(00)00424-3. No abstract available. PMID 11050365
- [Background] Saravanakumar K, Harvey A. Lumbar Zygapophyseal (Facet) Joint Pain. Rev Pain. 2008 Sep;2(1):8-13. doi: 10.1177/204946370800200103. PMID 26525677
- [Background] Scott D, Jull G, Sterling M. Widespread sensory hypersensitivity is a feature of chronic whiplash-associated disorder but not chronic idiopathic neck pain. Clin J Pain. 2005 Mar-Apr;21(2):175-81. doi: 10.1097/00002508-200503000-00009. PMID 15722811
- [Background] Seal RP, Wang X, Guan Y, Raja SN, Woodbury CJ, Basbaum AI, Edwards RH. Injury-induced mechanical hypersensitivity requires C-low threshold mechanoreceptors. Nature. 2009 Dec 3;462(7273):651-5. doi: 10.1038/nature08505. Epub 2009 Nov 15. PMID 19915548
- [Background] Smith HP, McWhorter JM, Challa VR. Radiofrequency neurolysis in a clinical model. Neuropathological correlation. J Neurosurg. 1981 Aug;55(2):246-53. doi: 10.3171/jns.1981.55.2.0246. PMID 7252548
- [Background] Solbiati L, Goldberg SN, Ierace T, Livraghi T, Meloni F, Dellanoce M, Sironi S, Gazelle GS. Hepatic metastases: percutaneous radio-frequency ablation with cooled-tip electrodes. Radiology. 1997 Nov;205(2):367-73. doi: 10.1148/radiology.205.2.9356616.
- [Background] Song KJ, Lee KB. Bilateral facet dislocation on L4-L5 without neurologic deficit. J Spinal Disord Tech. 2005 Oct;18(5):462-4. PMID 16189462
- [Background] Steele D, Baig KKK, Peter S. Evolving screening and surveillance techniques for Barrett's esophagus. World J Gastroenterol. 2019 May 7;25(17):2045-2057. doi: 10.3748/wjg.v25.i17.2045. PMID 31114132
- [Background] Suzuki H, Aono S, Inoue S, Imajo Y, Nishida N, Funaba M, Harada H, Mori A, Matsumoto M, Higuchi F, Nakagawa S, Tahara S, Ikeda S, Izumi H, Taguchi T, Ushida T, Sakai T. Clinically significant changes in pain along the Pain Intensity Numerical Rating Scale in patients with chronic low back pain. PLoS One. 2020 Mar 3;15(3):e0229228. doi: 10.1371/journal.pone.0229228. eCollection 2020. PMID 32126108
- [Background] Sweitzer SM, Colburn RW, Rutkowski M, DeLeo JA. Acute peripheral inflammation induces moderate glial activation and spinal IL-1beta expression that correlates with pain behavior in the rat. Brain Res. 1999 May 22;829(1-2):209-21. doi: 10.1016/s0006-8993(99)01326-8. PMID 10350552
- [Background] Tachihara H, Kikuchi S, Konno S, Sekiguchi M. Does facet joint inflammation induce radiculopathy?: an investigation using a rat model of lumbar facet joint inflammation. Spine (Phila Pa 1976). 2007 Feb 15;32(4):406-12. doi: 10.1097/01.brs.0000255094.08805.2f. PMID 17304129
- [Background] Twomey LT, Taylor JR, Taylor MM. Unsuspected damage to lumbar zygapophyseal (facet) joints after motor-vehicle accidents. Med J Aust. 1989 Aug 21;151(4):210-2, 215-7. doi: 10.5694/j.1326-5377.1989.tb115992.x. PMID 2761463
- [Background] Underwood MR, Dawes P. Inflammatory back pain in primary care. Br J Rheumatol. 1995 Nov;34(11):1074-7. doi: 10.1093/rheumatology/34.11.1074. PMID 8542211
- [Background] Van Boxem K, Huntoon M, Van Zundert J, Patijn J, van Kleef M, Joosten EA. Pulsed radiofrequency: a review of the basic science as applied to the pathophysiology of radicular pain: a call for clinical translation. Reg Anesth Pain Med. 2014 Mar-Apr;39(2):149-59. doi: 10.1097/AAP.0000000000000063. PMID 24553305
- [Background] Van Zundert J, de Louw AJ, Joosten EA, Kessels AG, Honig W, Dederen PJ, Veening JG, Vles JS, van Kleef M. Pulsed and continuous radiofrequency current adjacent to the cervical dorsal root ganglion of the rat induces late cellular activity in the dorsal horn. Anesthesiology. 2005 Jan;102(1):125-31. doi: 10.1097/00000542-200501000-00021. PMID 15618796
- [Background] Vatansever D, Tekin I, Tuglu I, Erbuyun K, Ok G. A comparison of the neuroablative effects of conventional and pulsed radiofrequency techniques. Clin J Pain. 2008 Oct;24(8):717-24. doi: 10.1097/AJP.0b013e318173c27a. PMID 18806537
- [Background] Velazquez KT, Mohammad H, Sweitzer SM. Protein kinase C in pain: involvement of multiple isoforms. Pharmacol Res. 2007 Jun;55(6):578-89. doi: 10.1016/j.phrs.2007.04.006. Epub 2007 Apr 29. PMID 17548207
- [Background] Veras del Monte LM, Bago J. Traumatic lumbosacral dislocation. Spine (Phila Pa 1976). 2000 Mar 15;25(6):756-9. doi: 10.1097/00007632-200003150-00020. PMID 10752113
- [Background] Vos T, Flaxman AD, Naghavi M, Lozano R, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gosselin R, Grainger R, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Ma J, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Years lived with disability (YLDs) for 1160 sequelae of 289 diseases and injuries 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2163-96. doi: 10.1016/S0140-6736(12)61729-2. PMID 23245607
- [Background] Verlaan JJ, Oner FC, Dhert WJ, Verbout AJ. Traumatic lumbosacral dislocation: case report. Spine (Phila Pa 1976). 2001 Sep 1;26(17):1942-4. doi: 10.1097/00007632-200109010-00026. PMID 11568711
- [Background] Walker K, Bowes M, Panesar M, Davis A, Gentry C, Kesingland A, Gasparini F, Spooren W, Stoehr N, Pagano A, Flor PJ, Vranesic I, Lingenhoehl K, Johnson EC, Varney M, Urban L, Kuhn R. Metabotropic glutamate receptor subtype 5 (mGlu5) and nociceptive function. I. Selective blockade of mGlu5 receptors in models of acute, persistent and chronic pain. Neuropharmacology. 2001;40(1):1-9. doi: 10.1016/s0028-3908(00)00113-1. PMID 11077065
- [Background] Watkins LR, Maier SF, Goehler LE. Immune activation: the role of pro-inflammatory cytokines in inflammation, illness responses and pathological pain states. Pain. 1995 Dec;63(3):289-302. doi: 10.1016/0304-3959(95)00186-7. PMID 8719529
- [Background] Weisshaar CL, Dong L, Bowman AS, Perez FM, Guarino BB, Sweitzer SM, Winkelstein BA. Metabotropic glutamate receptor-5 and protein kinase C-epsilon increase in dorsal root ganglion neurons and spinal glial activation in an adolescent rat model of painful neck injury. J Neurotrauma. 2010 Dec;27(12):2261-71. doi: 10.1089/neu.2010.1460. PMID 20925479
- [Background] Wilde VE, Ford JJ, McMeeken JM. Indicators of lumbar zygapophyseal joint pain: survey of an expert panel with the Delphi technique. Phys Ther. 2007 Oct;87(10):1348-61. doi: 10.2522/ptj.20060329. Epub 2007 Aug 7. PMID 17684091
- [Background] Willburger RE, Wittenberg RH. Prostaglandin release from lumbar disc and facet joint tissue. Spine (Phila Pa 1976). 1994 Sep 15;19(18):2068-70. doi: 10.1097/00007632-199409150-00011. PMID 7825047
- [Background] Winkelstein BA, Rutkowski MD, Sweitzer SM, Pahl JL, DeLeo JA. Nerve injury proximal or distal to the DRG induces similar spinal glial activation and selective cytokine expression but differential behavioral responses to pharmacologic treatment. J Comp Neurol. 2001 Oct 15;439(2):127-39. PMID 11596043
- [Background] Xu GY, Zhao ZQ. Change in excitability and phenotype of substance P and its receptor in cat Abeta sensory neurons following peripheral inflammation. Brain Res. 2001 Dec 27;923(1-2):112-9. doi: 10.1016/s0006-8993(01)03203-6. PMID 11743978
- [Background] Yamashita T, Minaki Y, Oota I, Yokogushi K, Ishii S. Mechanosensitive afferent units in the lumbar intervertebral disc and adjacent muscle. Spine (Phila Pa 1976). 1993 Nov;18(15):2252-6. doi: 10.1097/00007632-199311000-00018. PMID 8278841
- [Background] Yarmolenko PS, Moon EJ, Landon C, Manzoor A, Hochman DW, Viglianti BL, Dewhirst MW. Thresholds for thermal damage to normal tissues: an update. Int J Hyperthermia. 2011;27(4):320-43. doi: 10.3109/02656736.2010.534527. PMID 21591897